CLINICAL TRIAL: NCT00348777
Title: Evaluation of the Effects of a Water Cure on Gonarthrosis: Randomized Clinical Study Including Water Cure Versus Continuation of the Usual Treatment
Brief Title: THERMARTHROSE: Gonarthrosis and Water Cure
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Association Francaise pour la Recherche Thermale (Other)
Responsible Party: Pr Roques Christian, Association Francaise pour la Recherche Thermale
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DCIC 06 06
Record Dates: First submitted 2006-07-04; First posted 2006-07-06 (Estimated); Last update posted 2011-06-22 (Estimated); Status verified 2011-06

CONDITIONS: Osteoarthritis, Knee; Pain
Keywords: Visual analogic Scale of pain; Womac indice; SF-36 quality of life; Hydrotherapy
MeSH Terms: conditions — Osteoarthritis, Knee; Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): group with 18 days thermal cure
  Interventions: Drug: thermal cure
- 2 (Sham Comparator): group with no thermal cure but only access 3 days to watering place 6 months after inclusion
  Interventions: Drug: 3 days access to watering place at 6 months

INTERVENTIONS:
Drug: thermal cure — thermal cure of 18 days including movement in swimming pool, mud-bath, shower, massage and thermal steam
  Arms: 1
Drug: 3 days access to watering place at 6 months — access to watering place for movement in swimming pool, sauna and hammam.
  Arms: 2

SUMMARY:
The main objective of this study is to evaluate the therapeutic effect of a thermal treatment on gonarthrosis, with an increase of the number of patients presenting a clinically significant improvement.

DETAILED DESCRIPTION:
Gonarthrosis is a frequent pathology and the prevalence increase with age (prevalence: 6,1% in an adult population more than 30 years old and 40% after 75 years). It has a large impact on the quotidian life of the patients and it cause important costs for social protection. Relative to the treatment, numerous recommendations have been proposed (EULAR, ACR specifically). But no one of them recommends thermal treatment even if it is largely used in Europe and especially in France for the treatment of this pathology. Several prospective controlled randomized studies have evaluated the effect of the thermal treatments in rheumatology and some of them are relative, in part, to Gonarthrosis. So, we conduct a phase III randomized, controlled, single blind study evaluating the therapeutic effect at 6 month of a thermal cure on gonarthrosis.

In a situation of physical treatment, it's impossible to use a placebo as control: blind can't be respected. Whatever the methodology employed, non blind of the patient create a bias. So, we hope that the Zelen method for randomization will reduce the bias due to the dissatisfaction of the patients in the control group.

ELIGIBILITY:
Inclusion Criteria:

* ACR criteria: knee pain and one of the tree following conditions: Age > 50 years, Morning stiffness< 30 minutes and articular crackling.
* osteophytes visible on knee radiography.
* knee radiography less than 3 years old: face, schuss, axial of kneecap cliché.
* Actual gonarthrosis intensity on Visual Analogic Scale > or = 30mm.

Exclusion Criteria:

* arthrosis limited to the femoro-patellar compartments.
* severe depressive syndrome, psychosis.
* Thermal cure less than 6 month before.
* Contra-indication or predictable inability to tolerate thermal cure.
* Profession lied to hydrotherapy.
* previous knee treatments:

  * massage, physiotherapy and acupuncture since less than 1 month;
  * infiltration since less than 3 months;
  * NSAI since less than 5 days;
  * analgesic since less than 12 hours;
  * modification in the medicinal anti-arthrosis treatment since less than 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 462 (Actual)
Dates: Start 2006-06; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
the more small change clinically relevant of the WOMAC indice and/or of pain. | at 6 months

SECONDARY OUTCOMES:
WOMAC indice and pain (EVA) | at inclusion and 1, 3, 6 and 9 months
The clinically acceptable symptom for the patient | at 6 months
Clinical evaluation | at inclusion and 1, 3 and 6 months
Opinion of the patient and the physician | at 1, 3 and 6 months
Quality of life: questionnaire SF-36 | inclusion and 1, 3, 6 and 9 months
Treatments: medicinal consumption, physical treatments, hospitalization, consumption of cares getting back by the Medicaid of Savoie (CPAM, only for the study centre of Aix-les-Bains) | inclusion and 1,3,6 months

CONTACTS AND LOCATIONS:
Overall Officials: Romain FORESTIER, Dr, Principal Investigator — Président du Centre de Recherches Rhumatologiques et Thermales, Aix-les-Bains, France
Locations (3):
- France (3):
  - Cabinet médical, Balaruc-les-Bains
  - Cabinet Médical, Chambéry
  - Hôpital thermal, Dax

REFERENCES:
- [Background] Jordan KM, Arden NK, Doherty M, Bannwarth B, Bijlsma JW, Dieppe P, Gunther K, Hauselmann H, Herrero-Beaumont G, Kaklamanis P, Lohmander S, Leeb B, Lequesne M, Mazieres B, Martin-Mola E, Pavelka K, Pendleton A, Punzi L, Serni U, Swoboda B, Verbruggen G, Zimmerman-Gorska I, Dougados M; Standing Committee for International Clinical Studies Including Therapeutic Trials ESCISIT. EULAR Recommendations 2003: an evidence based approach to the management of knee osteoarthritis: Report of a Task Force of the Standing Committee for International Clinical Studies Including Therapeutic Trials (ESCISIT). Ann Rheum Dis. 2003 Dec;62(12):1145-55. doi: 10.1136/ard.2003.011742. PMID 14644851
- [Background] Ravaud P, Giraudeau B, Logeart I, Larguier JS, Rolland D, Treves R, Euller-Ziegler L, Bannwarth B, Dougados M. Management of osteoarthritis (OA) with an unsupervised home based exercise programme and/or patient administered assessment tools. A cluster randomised controlled trial with a 2x2 factorial design. Ann Rheum Dis. 2004 Jun;63(6):703-8. doi: 10.1136/ard.2003.009803. PMID 15140778
- [Background] Tubach F, Ravaud P, Baron G, Falissard B, Logeart I, Bellamy N, Bombardier C, Felson D, Hochberg M, van der Heijde D, Dougados M. Evaluation of clinically relevant changes in patient reported outcomes in knee and hip osteoarthritis: the minimal clinically important improvement. Ann Rheum Dis. 2005 Jan;64(1):29-33. doi: 10.1136/ard.2004.022905. Epub 2004 Jun 18. PMID 15208174
- [Background] Verhagen AP, de Vet HC, de Bie RA, Kessels AG, Boers M, Knipschild PG. Balneotherapy for rheumatoid arthritis and osteoarthritis. Cochrane Database Syst Rev. 2000;(2):CD000518. doi: 10.1002/14651858.CD000518. PMID 10796385
- [Background] Zelen M. Randomized consent designs for clinical trials: an update. Stat Med. 1990 Jun;9(6):645-56. doi: 10.1002/sim.4780090611. PMID 2218168
- [Derived] Forestier R, Genty C, Waller B, Francon A, Desfour H, Rolland C, Roques CF, Bosson JL. Crenobalneotherapy (spa therapy) in patients with knee and generalized osteoarthritis: a post-hoc subgroup analysis of a large multicentre randomized trial. Ann Phys Rehabil Med. 2014 Jun;57(4):213-27. doi: 10.1016/j.rehab.2014.03.001. Epub 2014 Mar 27. PMID 24745692
- [Derived] Forestier R, Desfour H, Tessier JM, Francon A, Foote AM, Genty C, Rolland C, Roques CF, Bosson JL. Spa therapy in the treatment of knee osteoarthritis: a large randomised multicentre trial. Ann Rheum Dis. 2010 Apr;69(4):660-5. doi: 10.1136/ard.2009.113209. Epub 2009 Sep 3. PMID 19734131